CLINICAL TRIAL: NCT00160446
Title: A Phase II Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of J867 Administered in Patients With Endometriosis
Brief Title: A Study to Evaluate the Safety and Effectiveness of Three Asoprisnil Doses in the Treatment of Women With Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Cynthia Mattia-Goldberg, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M99-110
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Endometriosis
Keywords: Pelvic pain; Dysmenorrhea; Dyspareunia; Infertility; Asoprisnil
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Dysmenorrhea; Dyspareunia; Infertility | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Asoprisnil
- 2 (Experimental)
  Interventions: Drug: Asoprisnil
- 3 (Experimental)
  Interventions: Drug: Asoprisnil
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil — 5mg Tablet, oral Daily for 12 weeks
  Arms: 1
Drug: Asoprisnil — 10 mg Tablet, oral Daily for 12 weeks
  Arms: 2
Drug: Asoprisnil — 25 mg Tablet, oral Daily for 12 weeks
  Arms: 3
Drug: Placebo — Tablet, oral Daily for 12 weeks
  Arms: 4

SUMMARY:
The objective of this study is to determine the safety and effectiveness of three doses of asoprisnil, compared to placebo, in the treatment of women with endometriosis.

DETAILED DESCRIPTION:
Endometriosis, the presence of endometrial tissue outside the uterus, is a progressive, estrogen-dependent disease that occurs in menstruating women of reproductive age. Although all major endometriosis therapies are effective for the treatment of pain, no single treatment is superior to others in terms of efficacy. The major drawbacks of the current medical therapies are severe side effects such as hot flushes and osteoporosis. The objective of this study is to determine the safety and efficacy of asoprisnil 5, 10, and 25 mg tablets, compared to placebo, administered daily for 12 weeks to women with endometriosis, by assessing whether asoprisnil administration diminishes the pelvic pain, dysmenorrhea, dyspareunia, excessive bleeding, and analgesic use associated with this disease and lessens the subjects' perceived pain symptoms. Otherwise healthy women with surgically confirmed endometriosis will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Surgically confirmed endometriosis
* History of menstrual cycles between 26 and 32 days
* Otherwise in good health
* Age 18-40 years, inclusive
* Subject had pain graded at Screening and Day 1 according to a scale suggested by Biberoglu and Berhman5 in at least one of the following categories:

  1. moderate or severe pelvic pain not related to menstruation, OR
  2. moderate or severe dysmenorrhea, OR
  3. moderate or severe pelvic tenderness elicited on pelvic examination accompanied by non-menstrual pelvic pain.
* Subject agrees to double barrier method of contraception

Exclusion Criteria:

* Any abnormal lab or procedure result the study-doctor considers important
* History of undiagnosed uterine bleeding or gynecological disorder
* Severe reaction(s) to hormone therapy
* History of osteoporosis or other metabolic bone disease
* Subject currently breast feeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2000-05; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Pain (dysmenorrhea, dyspareunia, pelvic pain) measured by daily diary | Mean change from baseline to Months 1, 2, 3

SECONDARY OUTCOMES:
Global efficacy question | Final visit
Pain (dysmenorrhea, dyspareunia, pelvic pain) pelvic tenderness and induration evaluated during office visits using modified Biberoglu and Behrman grading scale | Each monthly visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Abbott